CLINICAL TRIAL: NCT07404917
Title: The Effectiveness of Conservative Treatment With Added Kinesio Taping in Decreasing Pain and Improving Hand Function and Grip Strength Among Individuals With Lacertus Syndrome: A Pilot Randomized Controlled Trial
Brief Title: Kinesio Taping for Lacertus Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, Husam Taha, Principal Investigator, Arab American University (Palestine)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-2026/A/15/N
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Lacertus Syndrome
Keywords: Lacertus syndrome; Median nerve compression; Forearm pain; Kinesio Taping; Conservative treatment; Nerve gliding exercises; Rehabilitation; Feasibility study; Randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping Plus Conservative Treatment (Experimental): Participants in this arm will receive therapeutic Kinesio Taping applied with 25 to 50 percent stretch over the lacertus fibrosus region, reapplied every 2 to 3 days for 4 weeks. In addition, participants will receive the standardized conservative treatment protocol including patient education, median nerve gliding exercises, tendon gliding exercises, forearm stretching exercises, and activity modification guidelines.
  Interventions: Device: Kinesio Taping; Behavioral: Standardized Conservative Treatment
- Conservative Treatment Alone (Active Comparator): Participants in this arm will receive the standardized conservative treatment protocol alone, consisting of a 30-minute educational session about lacertus syndrome, a structured home exercise program (median nerve gliding exercises, tendon gliding exercises, and forearm muscle stretching performed twice daily), activity modification guidelines, and weekly telephone follow-up. All educational materials will be provided in Arabic.
  Interventions: Behavioral: Standardized Conservative Treatment

INTERVENTIONS:
Device: Kinesio Taping — Therapeutic elastic Kinesio Tape (5 cm width) applied with 25 to 50 percent stretch over the lacertus fibrosus in the proximal forearm. The tape is applied following standardized anatomical landmarks: anchor placed without stretch over the medial epicondyle region, therapeutic zone applied with stretch directly over the lacertus fibrosus, and terminal anchor placed without stretch over the proximal forearm. The initial application is performed by a trained therapist in the clinic. Participants are trained for home reapplication through hands-on demonstration, printed step-by-step instructions, and an instructional video. Tape is reapplied every 2 to 3 days for a total of 4 weeks. Adherence is monitored using tape application logs.
  Arms: Kinesio Taping Plus Conservative Treatment
Behavioral: Standardized Conservative Treatment — A 4-week standardized conservative treatment protocol consisting of four components: (1) Education: a 30-minute session covering lacertus syndrome anatomy and pathophysiology, activity modification guidelines, and ergonomic principles, with written materials provided in Arabic; (2) Exercise program: median nerve gliding exercises (3 sets of 10 repetitions, twice daily), tendon gliding exercises for flexor tendons (3 sets of 10 repetitions, twice daily), and forearm muscle stretching (30-second holds, 3 repetitions, twice daily), with access to an instructional video; (3) Activity modification: avoidance of repetitive pronation for more than 30 minutes continuously, regular breaks every 30 minutes during repetitive activities, use of ergonomic tools, and specific workplace modifications; (4) Follow-up: standardized weekly telephone check-ins to monitor compliance and address questions, with exercise logs for tracking adherence.

SUMMARY:
Background: Lacertus syndrome is a condition in which the median nerve is compressed at the lacertus fibrosus in the proximal forearm, leading to pain, numbness, weakness, and reduced hand function. The current standard treatment is surgical release. However, surgery may not be accessible or preferred by all patients, particularly in healthcare settings with limited resources. There is very little research on non-surgical treatment options for this condition.

Purpose: The purpose of this pilot study is to evaluate the feasibility and preliminary effectiveness of adding Kinesio Taping to a standardized conservative treatment program for adults diagnosed with lacertus syndrome.

Design: This is a single-blind, parallel-group, pilot randomized controlled trial. Thirty adults aged 18 to 65 years with a confirmed diagnosis of lacertus syndrome will be randomly assigned to one of two groups: (1) an experimental group receiving therapeutic Kinesio Taping applied over the lacertus fibrosus in addition to standardized conservative treatment, or (2) a control group receiving standardized conservative treatment alone. The conservative treatment includes patient education, nerve gliding exercises, tendon gliding exercises, stretching, and activity modification. The intervention period is 4 weeks.

Outcomes: The primary outcomes are feasibility measures including recruitment rate, retention rate, and adherence to the Kinesio Taping protocol. Secondary outcomes include pain intensity measured by the Numeric Pain Rating Scale, upper extremity function measured by the Quick Disabilities of the Arm, Shoulder and Hand questionnaire, grip strength measured by a hydraulic hand dynamometer, and pinch strength measured by a calibrated pinch gauge. All secondary outcomes are assessed at baseline and at 4 weeks.

Significance: This pilot study will provide essential data on the feasibility of conducting a Kinesio Taping intervention trial in the West Bank, Palestine, and will generate preliminary estimates of treatment effects to inform the design of a future definitive randomized controlled trial.

DETAILED DESCRIPTION:
Background and Rationale

Lacertus syndrome is a dynamic compression of the median nerve at the lacertus fibrosus (bicipital aponeurosis) in the proximal forearm. It is an increasingly recognized but often underdiagnosed cause of forearm pain, paresthesia, and functional disability. Up to 20% of patients presenting with signs of median nerve involvement may have compression at this level. The condition is frequently misdiagnosed as carpal tunnel syndrome or other nerve entrapment neuropathies due to overlapping clinical features.

Diagnosis relies on clinical examination including Hagert's triad (localized tenderness over the lacertus fibrosus, reproduction of symptoms with resisted forearm pronation, and reproduction of symptoms with resisted elbow flexion) and the Orthogonal Kinesiotaping Test (OKT), which has demonstrated 95% sensitivity and 89% specificity. Electrodiagnostic studies (electromyography and nerve conduction studies) are used to confirm median nerve involvement and exclude alternative diagnoses such as cervical radiculopathy.

Surgical release of the lacertus fibrosus is the current standard of care and has demonstrated high success rates. However, surgery may not be accessible, feasible, or preferred by all patients, particularly in resource-constrained healthcare systems. Despite this need, there is a critical gap in the evidence base for conservative management of lacertus syndrome. No high-quality randomized controlled trials have evaluated non-surgical interventions specifically designed for this condition.

Kinesio Taping is a therapeutic technique with a growing evidence base in musculoskeletal and neurological rehabilitation. Its proposed mechanisms of action include cutaneous mechanoreceptor stimulation, fascial decompression, proprioceptive enhancement, and neuromuscular re-education. Systematic reviews and meta-analyses have demonstrated that Kinesio Taping can reduce pain and improve function in carpal tunnel syndrome, another median nerve entrapment neuropathy, providing a rationale for investigating its application in lacertus syndrome.

Theoretical Framework

This study is guided by the International Classification of Functioning, Disability and Health (ICF) framework, specifically the Brief ICF Core Set for Hand Conditions. Within this framework, lacertus syndrome is conceptualized as a health condition leading to impairments in body functions (pain, muscle weakness, altered sensation) that affect activities (fine hand use, hand and arm use) and participation (self-care, domestic life, work). The Kinesio Taping intervention is positioned as a facilitator within the environmental factors domain. ICF codes targeted include b280, b730, b265, d440, d445, d5, d6, and d8.

Study Design and Randomization

This is a pilot, single-blind, parallel-group randomized controlled trial with a 1:1 allocation ratio, following SPIRIT 2013 guidelines and reported according to the CONSORT extension for pilot and feasibility trials.

Participants are allocated using a covariate-adaptive minimization procedure (Pocock and Simon method) implemented through validated randomization software. The algorithm balances age (40 years or younger versus older than 40), gender, symptom duration (4 to 12 weeks versus more than 12 weeks), baseline pain intensity (Numeric Pain Rating Scale score of 5 or less versus greater than 5), and recruitment site. A biased coin probability of 0.75 favors the allocation that minimizes imbalance while maintaining adequate randomness. The randomization sequence is generated and maintained by an independent statistician, with allocation concealment ensured through a secure, password-protected web-based system. The outcome assessor is blinded to group allocation; participants are instructed to wear long sleeves during assessments and to avoid discussing their treatment with the assessor.

Interventions

Experimental Group: Therapeutic Kinesio Taping applied with 25 to 50 percent stretch over the lacertus fibrosus region using 5-centimeter-width elastic therapeutic tape, following standardized anatomical landmarks (biceps tendon/lacertus fibrosus region, proximal pronator teres, and medial forearm fascia). The initial application is performed by a trained therapist; participants are then trained for home reapplication through hands-on demonstration, printed instructions, and an instructional video. Tape is reapplied every 2 to 3 days for 4 weeks, with adherence monitored using tape application logs. This group also receives the standardized conservative treatment described below.

Control Group: A standardized conservative treatment protocol consisting of a 30-minute educational session (anatomy, pathophysiology, activity modification, and ergonomic principles), a structured home exercise program (median nerve gliding exercises, tendon gliding exercises, and forearm muscle stretching, each performed twice daily), activity modification guidelines (including avoidance of sustained repetitive pronation and scheduled breaks during repetitive tasks), and weekly telephone follow-up. All materials are provided in Arabic.

Both groups receive the conservative treatment, ensuring that any observed differences are attributable to the addition of Kinesio Taping.

Data Analysis

Descriptive statistics will summarize feasibility outcomes and baseline characteristics. For secondary effectiveness outcomes, analysis follows the intention-to-treat principle. Change scores from baseline to 4 weeks will be compared between groups using independent t-tests or Mann-Whitney U tests depending on data distribution (assessed by the Shapiro-Wilk test). Effect sizes (Cohen's d) with 95% confidence intervals will be calculated. A significance level of 0.05 will be used. Multiple imputation with 20 imputed datasets will handle missing data, with sensitivity analyses including complete case analysis, per-protocol analysis, and pattern mixture models.

Safety Monitoring

All participants undergo skin patch testing prior to the first tape application. Adverse skin reactions are classified using a standardized four-grade scale and managed per a predefined protocol. Participants perform daily self-monitoring, with weekly clinical assessments by research staff. All adverse events are documented and reported to the Institutional Review Board according to Good Clinical Practice guidelines.

Ethical Considerations

This study is conducted in accordance with the Declaration of Helsinki and has been approved by the Institutional Review Board of the Arab American University of Palestine - Ramallah (approval number R-2026/A/15/N, approved February 3, 2026).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Confirmed clinical diagnosis of lacertus syndrome established by a physician specializing in orthopedics, physical medicine, or neurology following a standardized multi-modal diagnostic protocol
* Positive Hagert's triad, defined as the presence of all three of the following: (1) localized tenderness upon palpation of the lacertus fibrosus, (2) reproduction of symptoms during resisted forearm pronation, and (3) reproduction of symptoms during resisted elbow flexion
* Positive Orthogonal Kinesiotaping Test (OKT) conducted by a trained examiner
* Neurological evaluation excluding other median nerve entrapment syndromes such as carpal tunnel syndrome
* Electrodiagnostic studies (electromyography and nerve conduction studies) confirming median nerve involvement and ruling out alternative sources of neural compromise including cervical radiculopathy
* Symptom duration of at least 4 weeks to ensure subacute to chronic presentation
* Willing and able to provide written informed consent
* Able to attend all scheduled study visits and follow the home treatment protocol

Exclusion Criteria:

* Previous surgery for lacertus syndrome or any other median nerve entrapment condition in the affected arm
* Known allergy to Kinesio tape or adhesive materials
* Dermatological condition at the intended site of tape application (e.g., open wounds, active skin infection, eczema, psoriasis)
* Neurological disorder that could confound the assessment of lacertus syndrome symptoms (e.g., multiple sclerosis, diabetic peripheral neuropathy, cervical radiculopathy)
* Musculoskeletal disorder in the affected upper extremity that could confound symptom assessment (e.g., lateral or medial epicondylitis, shoulder impingement, rheumatoid arthritis affecting the hand or wrist)
* Current pregnancy
* Receipt of corticosteroid injection for lacertus syndrome within the past 3 months
* Current use of other therapeutic taping on the affected arm
* Cognitive impairment that would prevent understanding of study procedures or self-application of Kinesio tape

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Retention Rate | 4 weeks after baseline
  The proportion of randomized participants who complete the full 4-week intervention period and the final outcome assessment. Calculated as the number of participants completing the study divided by the total number of randomized participants, expressed as a percentage.
Recruitment Rate | Through study completion, approximately 6 months
  The number of eligible participants successfully enrolled into the study per month during the 6-month recruitment period. This will be calculated as the total number of randomized participants divided by the number of months of active recruitment.
Adherence Rate to Kinesio Taping Protocol | 4 weeks after baseline
  The proportion of prescribed Kinesio Tape applications that were completed by participants in the experimental group, as documented in standardized tape application logs. Calculated as the number of actual tape applications divided by the number of expected applications over the 4-week intervention period, expressed as a percentage.

SECONDARY OUTCOMES:
Change in Pain Intensity (Numeric Pain Rating Scale) | Baseline and 4 weeks
  Change in pain intensity from baseline to 4 weeks measured using the Numeric Pain Rating Scale (NRS). The NRS is an 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). A negative change score indicates improvement (pain reduction). The minimal clinically important difference is 2 points.
Change in Upper Extremity Function (QuickDASH) | Baseline and 4 weeks
  Change in upper extremity function from baseline to 4 weeks measured using the Quick Disabilities of the Arm, Shoulder and Hand questionnaire (QuickDASH), Arabic validated version. The QuickDASH is an 11-item questionnaire scored from 0 (no disability) to 100 (most severe disability). A negative change score indicates improvement (reduced disability). The minimal clinically important difference is 8 to 16 points.
Change in Grip Strength | Baseline and 4 weeks
  DescriptionChange in hand grip strength from baseline to 4 weeks measured using a calibrated hydraulic hand dynamometer following standardized protocols of the American Society of Hand Therapists. Measured in kilograms. The average of three trials with 30-second rest intervals will be recorded. A positive change score indicates improvement (increased strength)
Change in Tip Pinch Strength | Baseline and 4 weeks
  Change in tip pinch strength from baseline to 4 weeks measured using a calibrated pinch gauge following standardized protocols of the American Society of Hand Therapists. Measured in kilograms. The average of three trials with 30-second rest intervals will be recorded
Change in Key (Lateral) Pinch Strength | Baseline and 4 weeks
  Change in key (lateral) pinch strength from baseline to 4 weeks measured using a calibrated pinch gauge following standardized protocols of the American Society of Hand Therapists. Measured in kilograms. The average of three trials with 30-second rest intervals will be recorded.
Change in Palmar (Three-Jaw Chuck) Pinch Strength | Baseline and 4 weeks
  Change in palmar (three-jaw chuck) pinch strength from baseline to 4 weeks measured using a calibrated pinch gauge following standardized protocols of the American Society of Hand Therapists. Measured in kilograms. The average of three trials with 30-second rest intervals will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Elite for special orthopedic surgery, Ramallah, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article will be shared, after de-identification. This includes demographic characteristics, baseline and post-intervention scores for all outcome measures (Numeric Pain Rating Scale, QuickDASH, grip strength, and pinch strength), group allocation, and adherence data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months after publication of the main study results and available for 5 years following publication.
Access Criteria: Researchers who provide a methodologically sound proposal for use of the data. Proposals should be directed to the principal investigator (Husam Omar Taha) at the Arab American University of Palestine. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Ballestero-Perez R, Plaza-Manzano G, Urraca-Gesto A, Romo-Romo F, Atin-Arratibel MLA, Pecos-Martin D, Gallego-Izquierdo T, Romero-Franco N. Effectiveness of Nerve Gliding Exercises on Carpal Tunnel Syndrome: A Systematic Review. J Manipulative Physiol Ther. 2017 Jan;40(1):50-59. doi: 10.1016/j.jmpt.2016.10.004. Epub 2016 Nov 11. PMID 27842937
- [Background] Apard T, Ferembach B, Martinel V. Lacertus Syndrome Diagnosis With the Orthogonal Kinesiotaping Test. Plast Reconstr Surg Glob Open. 2025 Apr 23;13(4):e6728. doi: 10.1097/GOX.0000000000006728. eCollection 2025 Apr. PMID 40270558
- [Background] Hagert E. Clinical diagnosis and wide-awake surgical treatment of proximal median nerve entrapment at the elbow: a prospective study. Hand (N Y). 2013 Mar;8(1):41-6. doi: 10.1007/s11552-012-9483-4. PMID 24426891

DOCUMENTS (2):
  • Study Protocol (2026-02-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT07404917/Prot_000.pdf
  • Statistical Analysis Plan (2026-02-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT07404917/SAP_001.pdf